CLINICAL TRIAL: NCT00145795
Title: Randomized Trial of a Switch to a Kaletra + Current Dual Nucleoside Reverse Transcriptase Inhibitor (NRTI) Backbone Versus Continuation of the Current Regimen in Patients With Poor Immune Responses to Highly Active Antiretroviral Therapy (HAART) in Patients With Complete Viral Suppression: A Pilot Study
Brief Title: A Research Study to See if a Change in Therapy for HIV Infection Can Improve the Immune Response to Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11711B
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Results first posted 2013-08-27 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-05

CONDITIONS: HIV Infections
Keywords: HIV; HAART (Highly Active Anti-Retroviral Therapy) partial immune response; no immune response; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — lopinavir-ritonavir drug combination; Lopinavir; Ritonavir

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kaletra + Current Dual NRTI Backbone (Experimental): Patients in this arm received Kaletra in addition to their current Dual NRTI Backbone.
  Interventions: Drug: Kaletra + Current Dual NRTI Backbone
- Current Regimen (Active Comparator): Patients in this study arm continued their current regimen.
  Interventions: Drug: Current Regimen

INTERVENTIONS:
Drug: Kaletra + Current Dual NRTI Backbone
  Other Names: Lopinavir/ritonavir (LPV/r) + Current Dual NRTI Backbone
  Arms: Kaletra + Current Dual NRTI Backbone
Drug: Current Regimen
  Other Names: Current HIV treatment regimen
  Arms: Current Regimen

SUMMARY:
Our goal is to determine if a change in therapy to one containing Kaletra can improve the immune response in patients who have previously been immune partial responders or non-responders. We also are interested in knowing if this agent improves immune response by affecting cluster of differentiation 4 (CD4) + T cell death (apoptosis) or by further inhibiting (preventing) ongoing, low-level, viral replication to levels below detection by current viral load measurements. This will help us understand why immune responses to effective antiretroviral therapy are so different and help determine some possible guidelines for managing patients with poor immune responses.

Hypothesis: Patients with poor immune responses to HAART who receive Kaletra in place of their current PI or Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTIs) while continuing their current 2 NRTI backbone will have improved immune response to therapy compared to patients who continue their current regimen.

DETAILED DESCRIPTION:
To our knowledge our study is the first study showing persistent apoptosis in a subgroup of patients with complete viral suppression in association with poor immune recovery. Immune alterations independent of active viral replication may be responsible. Recent data suggests that immune responses to antiretroviral therapy depend on residual or restored thymic function. Improved CD4+ counts in patients despite virologic treatment failure are associated with greater thymic function, while poor T cell responses despite suppression of HIV are seen with decreased thymic function. Discordant immune responses may also be due to differential effects of particular antiretroviral agents on T cell apoptosis independent of viral suppression. For example, protease inhibitors have been shown to decrease rates of apoptosis of uninfected T cells. Viral replication is never completely suppressed with HAART, even when patients have undetectable plasma HIV RNA. Therefore, varying degrees of low level viral replication or replication in certain cellular compartments may continue to drive T cell apoptosis. Finally, our data suggests that ex vivo rates of Peripheral blood mononuclear cell (PBMC) apoptosis could potentially be used predict immune recovery or identify subgroups of patients who may benefit most from changes in HAART or adjunctive immunomodulatory therapies.

At this time, although there are excellent guidelines for how to evaluate and change therapy for patients with virologic failure, there are no recommendation and little data on approaches or strategies to change therapy for patients with poor immune responses. Kaletra (lopinavir/ritonavir) may be of benefit to patients with poor immune responses to HAART despite viral suppression. Kaletra may have greater potency and better suppression of viral replication that is below the level of detection by plasma polymerase chain reaction (PCR) for HIV-1 RNA. Kaletra also has an excellent pharmacokinetic profile which may result in superior inhibition of T cell apoptosis in vivo.

ELIGIBILITY:
Inclusion Criteria:

* HIV Infection documented CD4+ count within the last 30 days (or drawn with screening labs)
* Currently on a stable 3-drug HAART regimen including 2 NRTIs for > 6 month viral load (VL) < 50/mm3 for > 6 months, last within the last 30 days (or drawn with screening labs)
* Partial immune responder or immune non-responder
* Age > 18 years
* Labs (drawn at screening)
* Alanine transaminase (ALT) < 5 X the upper limit of normal (ULN)
* Total bili < 2 X ULN
* Creatinine < 2.0 mg/dL

Exclusion Criteria:

* Prior therapy with Kaletra
* Known hypersensitivity to Ritonavir
* Therapy the drugs with potential serious drug interactions: flecainide, propafenone, astemizole, terfenadine, rifampin, dihydroergotamine, ergonovine, ergotamine, methylergonovine, cisapride, pimozide, lovastatin, simvastatin, midazolam, triazolam, and St. John's wart.
* Pregnancy; breast feeding
* Current malignancy requiring CT
* Use of systemic corticosteroids, immunosuppressive, or cytotoxic agents within the last 45 days
* Fever and/or evidence of an active infectious complication
* Currently in another interventional clinical trial
* Receiving Interleukin-2 (IL-2) or any other cytokine or growth factor
* Enrollment in another interventional clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-04; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Pitrak, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Result] Pitrak DL, Estes R, Novak RM, Linnares-Diaz M, Tschampa JM. Beneficial effects of a switch to a Lopinavir/ritonavir-containing regimen for patients with partial or no immune reconstitution with highly active antiretroviral therapy despite complete viral suppression. AIDS Res Hum Retroviruses. 2011 Jun;27(6):659-67. doi: 10.1089/aid.2010.0230. Epub 2010 Dec 16. PMID 21054216

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from the outpatient clinics at the University of Chicago and the University of Illinois, with approval from the Institutional Review Board at each institution.
Period: Overall Study
Arm/Group | Kaletra + Current Dual NRTI Backbone | Current Regimen
Started | 10 | 10
Completed | 9 (1 patient discontinued early due to grade II gastrointestinal symptoms.) | 10
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kaletra + Current Dual NRTI Backbone | Current Regimen | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (14.4) | 40.5 (9.6) | 43 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 8 | 9 | 17
CD4 T cell count/mm^3 [Mean (Standard Deviation); unit: number of cells per cubic mm] | 172 (89) | 264 (106) | 218 (95.3)
Immune response at enrollment [Number; unit: participants] — We grouped patients according to their baseline absolute CD4+ lymphocyte counts before the initiation of HAART as follows: group 1, CD4+ <100/mm3; group 2, 100-199/mm3; group 3, 200-399/mm3, group 4, 400-699/mm3; and group 5, >= 700/mm3.
  Then, we categorized patients as complete or partial immune responders as follows. Complete immune responders have CD4+ counts increase to >700/mm3 after initiation of HAART. Partial immune responders have an increase in CD4+ count of >50% and improvement by at least one immunological grouping. All other patients are considered nonresponders.
  participants
    Nonresponder | 5 | 5 | 10
    Partial responder | 5 | 5 | 10
    Complete responder | 0 | 0 | 0
Duration of HAART prior to study entry [Mean (Standard Deviation); unit: months] | 28.8 (23.4) | 38.3 (28.8) | 33.6 (25.5)
HAART regimen at enrollment [Number; unit: participants] — NRTI: nucleoside reverse transcriptase inhibitor; NNRTI: non-nucleoside reverse transcriptase inhibitor; PI: protease inhibitor; Boosted PI: Combine low-dose ritonavir with a second PI and two or more NRTIs
  participants
    Two NRTIs + NNRTI | 7 | 6 | 13
    Two NRTIs + PI | 2 | 1 | 3
    Two NRTIs + boosted PI | 0 | 1 | 1
    Three NRTIs | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Immune Reconstitution [3 Months]
Description: Immune reconstitution is defined as the absolute CD4+ lymphocyte count after 3 months of therapy. Absolute CD4+ T cell count, our measure of immune recovery, was assessed in the clinical laboratory using fluorescent labeled monoclonal antibodies to the CD4 on lymphocytes. This is the main target cell for HIV infection. The absolute CD4+ T cell count is also the only clinically validated surrogate marker of immune dysfunction in HIV. CD4+ count is also our best predictor of morbidity and mortality outcomes.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: cells per cubic millimeter
Arm/Group | Kaletra + Current Dual NRTI Backbone | Current Regimen
Number analyzed (Participants) | 9 | 10
cells per cubic millimeter | 41.56 (34.84) | 49.40 (92.41)
Statistical Analysis 1: Comparison: Kaletra + Current Dual NRTI Backbone vs Current Regimen; Two-sample Student's t-test was used to examine the significance of the difference in mean absolute increase in CD4+ count at 3 months. Under the null hypothesis, CD4+ increase is similar for both treatment groups; Test type: Superiority or Other; p = 0.81, t-test, 2 sided — The significance level is 5%; This is a two-sample t-test assuming equal variances

2. Primary Outcome: Immune Reconstitution [6 Months]
Description: Immune reconstitution is defined as the absolute CD4+ lymphocyte count after 6 months of therapy. Absolute CD4+ T cell count, our measure of immune recovery, was assessed in the clinical laboratory using fluorescent labeled monoclonal antibodies to the CD4 on lymphocytes. This is the main target cell for HIV infection. The absolute CD4+ T cell count is also the only clinically validated surrogate marker of immune dysfunction in HIV. CD4+ count is also our best predictor of morbidity and mortality outcomes.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: cells per cubic millimeter
Arm/Group | Kaletra + Current Dual NRTI Backbone | Current Regimen
Number analyzed (Participants) | 9 | 10
cells per cubic millimeter | 116 (108) | 32 (49)
Statistical Analysis 1: Comparison: Kaletra + Current Dual NRTI Backbone vs Current Regimen; Two-sample Student's t-test was used to examine the significance of the difference in mean absolute increase in CD4+ count at 6 months. Under the null hypothesis, CD4+ increase is similar for both treatment groups; Test type: Superiority or Other; p = 0.03, t-test, 2 sided — Significance level is 5%; This is a two-sample t-test assuming equal variances

3. Secondary Outcome: Rates of ex Vivo T Cell Apoptosis: CD4+ Memory Cell Population [3 Months]
Description: Ex vivo T cell apoptosis can be assessed many different ways. The use of propidium iodide staining to determine the proportion of isolated cells that have undergone apoptosis after ex vivo incubation is a standard method that has been used by many investigators. Apoptotic cells intercalate less PI into their DNA, and on flow cytometry, this cell population is identified by a decrease in mean fluorescence (shift to the left). We have experience with this assay, and we have published on the use of method for determining rates of ex vivo apoptosis for different immune effector cells.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percent apoptosis
Arm/Group | Kaletra + Current Dual NRTI Backbone | Current Regimen
Number analyzed (Participants) | 9 | 10
percent apoptosis | 15.27 (6.99) | 24.53 (13.45)
Statistical Analysis 1: Comparison: Kaletra + Current Dual NRTI Backbone vs Current Regimen; Two-sample Student's t-test was used to assess the difference in mean percent apoptosis for the CD4+ memory cell population at 3 months. Under the null hypothesis, percent CD4+ memory cell apoptosis is similar for both treatment groups; Test type: Superiority or Other; p = 0.08, t-test, 2 sided — The significance level is 5%; This is a two-sample t-test assuming equal variances

4. Secondary Outcome: Rates of ex Vivo T Cell Apoptosis: CD4+ naïve Cell Population [3 Months]
Description: as for outcome 3
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percent apoptosis
Arm/Group | Kaletra + Current Dual NRTI Backbone | Current Regimen
Number analyzed (Participants) | 9 | 10
percent apoptosis | 16.60 (9.62) | 22.53 (13.35)
Statistical Analysis 1: Comparison: Kaletra + Current Dual NRTI Backbone vs Current Regimen; Two-sample Student's t-test was used to assess the difference in mean percent apoptosis for the CD4+ naïve cell population at 3 months. Under the null hypothesis, percent CD4+ naïve cell apoptosis is similar for both treatment groups; Test type: Superiority or Other; p = 0.29, t-test, 2 sided — The significance level is 5%; This is a two-sample t-test assuming equal variances

5. Secondary Outcome: Rates of ex Vivo T Cell Apoptosis: CD4+ Memory Cell Population [6 Months]
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percent apoptosis
Arm/Group | Kaletra + Current Dual NRTI Backbone | Current Regimen
Number analyzed (Participants) | 9 | 10
percent apoptosis | 14.10 (5.53) | 17.94 (9.20)
Statistical Analysis 1: Comparison: Kaletra + Current Dual NRTI Backbone vs Current Regimen; Two-sample Student's t-test was used to assess the difference in mean percent apoptosis for the CD4+ memory cell population at 6 months. Under the null hypothesis, percent CD4+ memory cell apoptosis is similar for both treatment groups; Test type: Superiority or Other; p = 0.29, t-test, 2 sided — The significance level is 5%; This is a two-sample t-test assuming equal variances

6. Secondary Outcome: Rates of ex Vivo T Cell Apoptosis: CD4+ naïve Cell Population [6 Months]
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percent apoptosis
Arm/Group | Kaletra + Current Dual NRTI Backbone | Current Regimen
Number analyzed (Participants) | 9 | 10
percent apoptosis | 10.03 (5.25) | 18.92 (10.65)
Statistical Analysis 1: Comparison: Kaletra + Current Dual NRTI Backbone vs Current Regimen; Two-sample Student's t-test was used to assess the difference in mean percent apoptosis for the CD4+ naïve cell population at 6 months. Under the null hypothesis, percent CD4+ naïve cell apoptosis is similar for both treatment groups; Test type: Superiority or Other; p = 0.04, t-test, 2 sided — The significance level is 5%; This is a two-sample t-test assuming equal variances

7. Secondary Outcome: Rates of ex Vivo T Cell Apoptosis: CD8+ Cell Population [3 Months]
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percent apoptosis
Arm/Group | Kaletra + Current Dual NRTI Backbone | Current Regimen
Number analyzed (Participants) | 9 | 10
percent apoptosis | 20.92 (6.63) | 16.74 (7.15)
Statistical Analysis 1: Comparison: Kaletra + Current Dual NRTI Backbone vs Current Regimen; Two-sample Student's t-test was used to assess the difference in mean percent apoptosis for the CD8+ cell population at 3 months. Under the null hypothesis, percent CD8+ cell apoptosis is similar for both treatment groups; Test type: Superiority or Other; p = 0.21, t-test, 2 sided — The significance level is 5%; This is a two-sample t-test assuming equal variances

8. Secondary Outcome: Rates of ex Vivo T Cell Apoptosis: CD8+ Cell Population [6 Months]
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percent apoptosis
Arm/Group | Kaletra + Current Dual NRTI Backbone | Current Regimen
Number analyzed (Participants) | 9 | 10
percent apoptosis | 17.07 (9.38) | 19.01 (6.99)
Statistical Analysis 1: Comparison: Kaletra + Current Dual NRTI Backbone vs Current Regimen; Two-sample Student's t-test was used to assess the difference in mean percent apoptosis for the CD8+ cell population at 6 months. Under the null hypothesis, percent CD8+ cell apoptosis is similar for both treatment groups; Test type: Superiority or Other; p = 0.61, t-test, 2 sided — The significance level is 5%; This is a two-sample t-test assuming equal variances

9. Secondary Outcome: Clinical HIV-related Events
Description: Number of participants experiencing clinical HIV-related events as defined by category A, category B, and Appendix B in the "1993 Revised Classification System for HIV Infection and Expanded Surveillance Case Definition for AIDS Among Adolescents and Adults" (http://www.cdc.gov/mmwr/preview/mmwrhtml/00018871.htm).
Time Frame: 6 months
Measure: Number; unit: number of participants with event(s)
Arm/Group | Kaletra + Current Dual NRTI Backbone | Current Regimen
Number analyzed (Participants) | 9 | 10
number of participants with event(s) | 0 | 0

10. Secondary Outcome: Rates of Virologic Failure
Description: Virologic failure defined as HIV RNA > 2,000 copies/mL
Time Frame: 6 months
Measure: Number; unit: percentage of randomized subjects
Arm/Group | Kaletra + Current Dual NRTI Backbone | Current Regimen
Number analyzed (Participants) | 9 | 10
percentage of randomized subjects | 0 | 0

ADVERSE EVENTS:
Time Frame: 0-6 months
Arm/Group | Kaletra + Current Dual NRTI Backbone | Current Regimen
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Kaletra + Current Dual NRTI Backbone (N=10) | Current Regimen (N=10)
Nausea dyspepsia (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes